CLINICAL TRIAL: NCT03586544
Title: Asthma and Childhood Obesity: Understanding Potential Mechanisms and Identifying Strategies to Improve Respiratory Symptoms
Brief Title: Reducing Exercise-induced Bronchoconstriction in Children With Asthma and Obesity
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was halted prematurely due to COVID 19.
Sponsor: University of Nevada, Las Vegas (Other)
Responsible Party: Principal Investigator, Dharini M Bhammar, Assistant Professor, University of Nevada, Las Vegas
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 1131374-2
Record Dates: First submitted 2018-07-02; First posted 2018-07-13 (Actual); Results first posted 2021-07-21 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Asthma in Children; Obesity, Childhood; Exercise Induced Bronchospasm
Keywords: pediatric; bronchoconstriction
MeSH Terms: conditions — Pediatric Obesity; Asthma, Exercise-Induced | interventions — Albuterol

STUDY DESIGN:
Intervention Model Description: 2x3 mixed ANOVA. 2 between groups: children with and without obesity. 3 within groups: control, interval warm-up, pretreatment with bronchodilator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Albuterol first (Experimental): Order albuterol and then interval warm up (IWU)
  Interventions: Drug: Albuterol Sulfate; Behavioral: Interval Warm-up exercise
- Interval warm-up first (Experimental): Order is interval warm up (IWU) and then albuterol
  Interventions: Drug: Albuterol Sulfate; Behavioral: Interval Warm-up exercise

INTERVENTIONS:
Drug: Albuterol Sulfate — Participants will inhale 2 puffs of albuterol (90mcg per actuation). After 15 minutes, participants will undergo an exercise induced bronchoconstriction test
  Other Names: Ventolin
Behavioral: Interval Warm-up exercise — Participants will undergo eight 30 sec bouts of high intensity exercise with 45 second recovery between bouts. After 15 minutes, participants will undergo an exercise induced bronchoconstriction test

SUMMARY:
Guidelines from the American Thoracic Society strongly recommend interval warm-up exercise before planned exercise to reduce exercise-induced bronchoconstriction severity. However, no empirical data on the effects of interval warm-up exercise on exercise-induced bronchoconstriction severity are available in obese asthmatic children, where excess fat exerts such an unfavorable burden on the respiratory system, particularly during exercise. The objective of this study is to investigate the effects of interval warm-up exercise on exercise-induced bronchoconstriction severity in obese and nonobese asthmatic children. Our approach will be to investigate exercise tolerance, respiratory function, and exercise-induced bronchoconstriction severity and the effects of (1) 8x30sec interval warm-up & (2) pretreatment with a bronchodilator compared with a no-treatment control on exercise-induced bronchoconstriction severity in 8-12 yr, prepubescent, obese and nonobese asthmatic children.

[Aim]: To investigate the effects of interval warm-up exercise on exercise-induced bronchoconstriction severity. [Hypothesis]: Interval warm-up exercise will reduce exercise-induced bronchoconstriction severity after an exercise challenge test to a similar extent as bronchodilator and better than control.

DETAILED DESCRIPTION:
Note related to early termination: Although the intent of the study was to compare obese and nonobese children, early termination precluded us from completing this analysis and thus the pooled results are included in the results. The brief summary has been updated to reflect the presented results.

The investigators will enroll prepubescent, 8 - 12 yr old, obese (body mass index > 95th percentile; N=25) and nonobese (body mass between 16th and 84th percentile; N=25) children with mild asthma. The investigators will investigate the severity of exercise-induced bronchoconstriction during planned exercise performed 15 minutes after the following three conditions performed on separate days in a random order: (1) 8x30sec interval warm-up, (2) short-acting beta agonist or albuterol, & (3) control, in prepubescent, 8 - 12 yr old, obese and nonobese children with mild asthma.

The investigators will measure the following in all participants:

1. Pulmonary function: spirometry, lung volumes, diffusing capacity of lung for carbon monoxide, maximum voluntary ventilation, maximal inspiratory and expiratory pressures, airway resistance, and expired nitric oxide
2. Exercise tolerance during graded cycle ergometry: Gas exchange, ventilation, heart rate, blood pressure, pulse oximetry, electrocardiogram
3. Ratings of perceived breathlessness and exercise induced bronchoconstriction in response to a 6 minute high-intensity exercise challenge after three conditions performed on three separate days:

Three conditions that will precede the exercise challenge include:

1. 8x30sec of interval warm-up 15min prior to exercise challenge: This includes eight 30sec bouts of high-intensity interval exercise at 85-95% of HRmax, with 45sec of recovery between.
2. Two puffs of albuterol 15 min prior to exercise challenge
3. Control: seated rest for 15min prior to exercise challenge

Control visit was always completed first. The order of the albuterol and interval warm-up exercise visits was randomized.

ELIGIBILITY:
Inclusion Criteria:

* no history of smoking, no history or evidence of heart disease, no history of uncontrolled hypertension, no documented and/or diagnosed sleep disorders, no diagnosed diabetes, no metabolic disorders, no history of significant mental illness, no dietary restrictions, no serious health conditions, or no musculoskeletal abnormality that would preclude exercise.
* Normal weight children with a body mass index between the 16th and 84th percentile
* Obese children with a body mass index > 95th percentile but less than 170% above the 95th percentile and less than an absolute body mass index of 40 kg·m2
* Pulmonary function criteria 1) forced vital capacity ≥ 80% predicted, 2) forced expiratory volume in the first second (FEV1) ≥ 75% predicted, and total lung capacity ≥ 80% predicted

Exclusion Criteria:

* Children with significant diseases other than obesity and mild asthma will be excluded. A significant disease is defined as either a disease that in the opinion of the PI or medical consultant Dr. Craig Nakamura may put the participant at risk because of participation in the study or a disease that may influence the results of the study or the patient's ability to participate in the study.
* Children who cannot follow directions (e.g., eating before testing), adequately perform procedures (e.g., pulmonary function tests), or keep appointments (e.g., no shows for testing), will be excluded from study participation.
* Because the risk of severe exercise induced bronchoconstriction increases in children with moderate or severe obstructive airway disease, children with FEV1 < 75% predicted will be excluded from the study. Diagnosis of asthma (i.e., airway responsiveness with reversible obstruction) will be established by spirometry (i.e., improvement of FEV1 of ≥8% after administration of bronchodilator).
* Children without reversible airway obstruction will also be excluded from the study.
* Children who have been hospitalized for an asthma exacerbation or who have taken oral glucocorticoids for asthma in the past year, and children who have been admitted to an intensive care unit or been intubated because of their asthma in the past five years, will be excluded to reduce the risk of exacerbation during the study.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2021-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dharini M Bhammar, Ph.D., Principal Investigator — University of Nevada, Las Vegas
Locations (1):
- Childrens Lung Specialists, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No
There is no current plan to share individual participant data.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment:
  34 participants were screened for eligibility between 9/18/2018 - 3/13/2020. Participants were recruited from the Children's Lung Specialists Pediatric Pulmonology clinic.
Pre-assignment Details: 18 out of 34 enrolled participants were randomized. Of those not randomized (N=16), 10 did not meet inclusion criteria, 5 declined to participate, and 1 was not randomized because we terminated the study early. Of the 18 participants randomized, 2 did not complete all study visits: 1 because they declined to continue and 1 because of leg pain during exercise.
Groups:
- Order 1: Albuterol First, Interval Warm-up Second: Participants first received albuterol on one day only. After at least 72 h, they completed the interval warm up on one day only. This was an acute study. There is no washout per se.
- Order 2: Interval Warm-up First, Albuterol Second: Participants first completed interval warm up exercise on one day only. After at least 72 h, they recieved the albuterol (180ug) on one day only. This was an acute study. There is no washout per se.
Period: First Intervention
Arm/Group | Order 1: Albuterol First, Interval Warm-up Second | Order 2: Interval Warm-up First, Albuterol Second
Started | 6 | 12
Completed | 6 | 11
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Second Intervention
Arm/Group | Order 1: Albuterol First, Interval Warm-up Second | Order 2: Interval Warm-up First, Albuterol Second
Started | 6 | 11
Completed | 6 | 10
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline analysis is shown for all randomized participants including the two participants who did not complete the interval warm-up first arm.
Groups:
- Albuterol First: Children will complete an exercise induced bronchoconstriction test preceded by: 1) Control, 2) pretreatment with 'Albuterol' and 3) interval warm-up exercise and
  Control visit was always completed first. The order of albuterol and interval warm-up was randomized. In this arm, albuterol visit was completed first.
- Interval Warm up First: Children will complete an exercise induced bronchoconstriction test preceded by: 1) Control, 2) pretreatment with 'Albuterol' and 3) interval warm-up exercise and
  Control visit was always completed first. The order of albuterol and interval warm-up was randomized. In this arm, interval warm-up visit was completed first.
- Total: Total of all reporting groups
Arm/Group | Albuterol First | Interval Warm up First | Total
Number analyzed (Participants) | 6 | 12 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.6 (0.9) | 10.4 (1.0) | 10.5 (0.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 2 | 10 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 10
  Not Hispanic or Latino | 2 | 6 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 4 | 10 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 6 | 12 | 18

OUTCOME MEASURES:

1. Primary Outcome: Maximum % Change in Forced Expiratory Volume in the First Second (FEV1)
Description: The change in FEV1 from before to after the exercise induced bronchoconstriction test.
  For the control condition, the change in FEV1 was measured from before the 6min exercise challenge test to up to 30 min after the exercise challenge test. The control condition was completed before participants were randomized to either albuterol or interval warm-up. This "control" condition is our reference condition because any improvement noted with albuterol or interval warm-up exercise should be compared against the control condition.
Time Frame: The change in FEV1 will be assessed for up to 30 minutes after completing the exercise induced bronchoconstriction test
Population: Two participants did not complete the interval warm-up arm and there results are not reported.
Measure: Mean (Standard Deviation); unit: percentage change
Groups:
- Albuterol First: Albuterol first and then interval warm up
- Interval Warm-up First: Interval warm-up first and then albuterol
Arm/Group | Albuterol First | Interval Warm-up First
Number analyzed (Participants) | 6 | 10
percentage change
  Control | 1.91 (7.47) | -0.84 (12.22)
  Albuterol | 7.98 (17.12) | 13.03 (6.72)
  Interval Warm up | 1.12 (14.90) | -1.72 (11.11)

ADVERSE EVENTS:
Time Frame: For our participants, the five visits were completed within 6.9 ± 2.4 weeks (Range: 3.6-11.1 weeks).
Groups:
- Albuterol Intervention: 180 ug of albuterol given on one day in this acute study.
- Interval Warm-up Intervention: Interval warm-up exercise completed on one day in this acute study.
Arm/Group | Albuterol Intervention | Interval Warm-up Intervention
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/18
Other Adverse Events (participants affected / at risk) | 0/16 | 2/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Albuterol Intervention (N=16) | Interval Warm-up Intervention (N=18)
Vocal cord dysfunction during exercise (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1/12 (1) — Complained of shortness of breath towards the end of the exercise challenge test on the day of the interval warm-up visit. Evaluated by pediatric pulmonologist. Resolved spontaneously. Patient taught sniff and blow technique for future.
Leg pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1/12 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-10): https://cdn.clinicaltrials.gov/large-docs/44/NCT03586544/Prot_SAP_004.pdf
  • Informed Consent Form (2020-12-11): https://cdn.clinicaltrials.gov/large-docs/44/NCT03586544/ICF_003.pdf